CLINICAL TRIAL: NCT01715779
Title: An Observational Follow-up Study of Patients Who Experienced Thromboembolic Events in the ENABLE Studies
Brief Title: Follow-up Study of Patients Who Experienced Thromboembolic Events in the ENABLE Studies
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 116951; WWE116951 (Other: GSK); EPI40685 (Other: GSK)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C
Keywords: Liver transplantation; ENABLE; observational; mortality; Thromboembolic Events; Hepatic decompensation; Long-Term follow-up; TEE
MeSH Terms: conditions — Hepatitis C; Thromboembolism | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who experienced a thromboembolic event: Patients who experienced a thromboembolic event during participation in the ENABLE clinical trials.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag exposure

SUMMARY:
The objective of this observational study is to characterize long-term (5 years post event) clinical outcomes in patients who experienced a thromboembolic event (TEE) during participation in the GSK ENABLE clinical trials.

Patients eligible for the study are patient who experienced a TEE during participation in the ENABLE trials. Each included patient will be followed for a period of 5 years from the date of their first TEE. Demographic and clinical characteristics will be collected for the index date (time of TEE) and every sixth month during the follow-up period, information will be collected for the outcomes of interests: mortality, new TEE, hepatic decompensation, evaluation for liver transplant and result of evaluation, and liver transplantation.

All information will collected by medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Patients with portal vein thrombosis (PVT)
* Patients with deep vein thrombosis (DVT)
* Patients with pulmonary embolism (PE)
* Patients with myocardial infarction (MI)
* Patients with unstable angina
* Patients with transient ischemic attack (TIA)
* Patients with ischemic stroke
* Patients with other TEE including embolism, thrombosis, phlebitis, and thrombophlebitis at other locations

Exclusion Criteria:

* There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients under study are patients who experienced a thromboembolic event during participation in the ENABLE clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Mortality. Patients who experience a thromboembolic event (TEE) and died during study participation. | The patients will be followed from 5 years from first occurrence of thromboembolic event.
  An observational study following patients who experienced a thromboembolic event (TEE) during participation in the ENABLE trials. Each included patient will be followed for a period of 5 years from the date of their first TEE. Demographic and clinical characteristics will be collected for the index date (time of TEE) and every sixth month during the follow-up period. All information will collected by medical record review.
New Thromboembolic Events (TEE). Patients who experienced a new TEE during participation. | The patients will be followed from 5 years from first occurrence of thromboembolic event.
  An observational study following patients who experienced a thromboembolic event (TEE) during participation in the ENABLE trials. Each included patient will be followed for a period of 5 years from the date of their first TEE. Demographic and clinical characteristics will be collected for the index date (time of TEE) and every sixth month during the follow-up period. All information will collected by medical record review.
Hepatic decompensation. Patients who experienced a hepatic decompensation during study participation. | The patients will be followed from 5 years from first occurrence of thromboembolic event.
  An observational study following patients who experienced a thromboembolic event (TEE) during participation in the ENABLE trials. Each included patient will be followed for a period of 5 years from the date of their first TEE. Demographic and clinical characteristics will be collected for the index date (time of TEE) and every sixth month during the follow-up period. All information will collected by medical record review.
Evaluation for liver transplant and result of evaluation. | The patients will be followed from 5 years from first occurrence of thromboembolic event.
  An observational study following patients who experienced a thromboembolic event (TEE) during participation in the ENABLE trials. Each included patient will be followed for a period of 5 years from the date of their first TEE. Demographic and clinical characteristics will be collected for the index date (time of TEE) and every sixth month during the follow-up period. All information will collected by medical record review.
Liver transplantation. Patients who experienced a Liver transplantation during study participation. | The patients will be followed from 5 years from first occurrence of thromboembolic event.
  An observational study following patients who experienced a thromboembolic event (TEE) during participation in the ENABLE trials. Each included patient will be followed for a period of 5 years from the date of their first TEE. Demographic and clinical characteristics will be collected for the index date (time of TEE) and every sixth month during the follow-up period. All information will collected by medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals